CLINICAL TRIAL: NCT03146949
Title: Does the Type of Oxygenator Influence Arterial Blood Concentration of Isoflurane During Cardiopulmonary Bypass?
Brief Title: Blood Isoflurane Concentration and the Oxygenator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AC16130
Record Dates: First submitted 2017-04-06; First posted 2017-05-10 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Cardiopulmonary Bypass

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Primary outcome assessor is masked. The primary outcome involves the analysis of blood concentrations of isoflurane, and the laboratory will not be given information on allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sorin Inspire Oxygenator (Active Comparator): Sorin Inspire Oxygenator is used on the cardiopulmonary bypass machine
  Interventions: Device: Sorin Inspire Oxygenator
- Medtronic Affinity Fusion Oxygenator (Active Comparator): Medtronic Affinity Fusion Oxygenator is used on the cardiopulmonary bypass machine
  Interventions: Device: Medtronic Affinity Fusion

INTERVENTIONS:
Device: Sorin Inspire Oxygenator — This is an oxygenator manufactured by the Sorin group. It is a hollow fibre polypropylene oxygenator.
  Arms: Sorin Inspire Oxygenator
Device: Medtronic Affinity Fusion — This is an oxygenator manufactured by the Medtronic group. It is a hollow fibre polypropylene oxygenator.
  Arms: Medtronic Affinity Fusion Oxygenator

SUMMARY:
This study compares two oxygenators commonly in use to establish whether they effect the amount of isoflurane in the patient's blood. Half of the patients will be placed in a group using the Sorin Inspire oxygenator and half into the group using the Medtronic Affinity Fusion oxygenator.

DETAILED DESCRIPTION:
Cardiopulmonary bypass (CPB) is the keystone of most of these surgeries, as it allows for the maintenance of patient circulation without the requirement for a beating heart or breathing lungs. However, in doing so, CPB creates a unique set of difficulties associated with administering and maintaining anaesthesia. Firstly, the usual route of administration of inhalational anaesthetics, such as isoflurane, via the lungs is impossible. Secondly, clinical signs used to assess depth of anaesthesia, such as heart rate and systemic arterial blood pressure, are obscured by the mechanical support of the circulation. As a consequence, maintaining and assessing the depth of anaesthesia achieved during CBP provides challenges for the anaesthetists.

One common approach to administering anaesthesia during CBP involves the delivery of an inhalational anaesthetic agent, such as isoflurane, into the sweep gas supply to the oxygenator. Whilst classic terminology describes agents such as isoflurane as inhalational, in CPB this may cause confusion due to the delivery of the agent through the oxygenator as opposed to the lungs. Therefore, the alternative name of volatile anaesthetic agents is utilised in this protocol. Isoflurane concentrations ranging between 1% and 2.5% have been used by several anaesthetists at the Royal Infirmary of Edinburgh (RIE) for many years. This pragmatic approach has been found to produce clinically adequate depth of anaesthesia when either of the two oxygenators in routine use at the RIE are employed. Indeed, it has been shown using an electro-encephalographic (EEG) technique of assessing depth of anaesthesia, known as the Bispectral Index (BIS), that administering 2.5% isoflurane produces a more than adequate depth of anaesthesia. However, as discussed below, the interpretation of this finding is limited by the profound effect of hypothermia, which is commonly induced on CPB, has on BIS.

BIS is frequently utilised by anaesthetists to monitor anaesthetic depth. It involves real-time monitoring brain electrical waves using an EEG to produce a dimensionless number between 0 (no cortical brain activity) and 100 (awake), with 40 to 60 being widely accepted as a score suitable for general anaesthesia. Whilst BIS is frequently used in practice, as it has been shown to reduce anaesthetic awareness and increase emergence time, it is not without controversy as there is conflicting evidence regarding its reliability, particularly during CPB as low body temperature is known to affect its readings.

Considering the limitations of BIS, other methods can be employed to estimate depth of anaesthesia. The arterial blood concentration of the volatile agent is a good surrogate, as the concentration of agent in the brain will equilibrate with that of the blood.

Whilst this measurement provides a definitive value of how much anaesthetic agent is reaching the brain, it is impractical for clinical use because of the long duration and complexity of laboratory analysis that is required. Therefore, another approach can use the concentration of the volatile agent in the gases exhausted from the oxygenator in order to estimate the arterial blood concentration. This approach is analogous to using the end-tidal concentration that is expired from the lungs during routine general anaesthesia. Oxygenator exhaust, unlike arterial blood concentration, would be practical in a clinical scenario as the oxygenator exhaust from CPB can be attached to a standard anaesthetic gas monitor. Indeed, there is evidence that suggests measuring the oxygenator exhaust concentration of volatile anaesthetic agent is a good surrogate of arterial blood levels.

The oxygenator acts as the key interface between the patient's blood and volatile anaesthetic agent, and their availability is essential for CPB to go ahead. The RIE stock and routinely use two makes of oxygenator in case of manufacture supply problems - in which event the perfusionist would be familiar with using both. Both oxygenators are membrane in nature, consisting of microporous polypropylene hollow fibres. One is the Medtronic Affinity Fusion ('Fusion') and the other is Sorin Inspire ('Inspire'), with the choice of which is used being at the discretion of the perfusionist. Both oxygenators possess a similar design, with the patient's blood flowing over the fibers and a mixture of air and oxygen passing through them, allowing for gas exchange to occur, and crucially allowing the passage of volatile anaesthetic agent into the patient's blood. As the manufacture and design of various oxygenators are different, each possesses a unique set of transfer characteristics, which has been shown in bench tests to affect the uptake and elimination of isoflurane. The combined experience of the anaesthetists at the RIE indicates there is no clinical difference between the two different oxygenators in routine use or the resulting anaesthesia, however these bench tests suggest there may be some difference in transfer characteristics which may be established by small differences measured in the arterial blood level of isoflurane.

It also follows that if there are differences in arterial blood levels, other methods of measuring depth of anaesthesia, such as BIS and oxygen exhaust concentration of anaesthetic agent, may also show differences dependent on the oxygenator used. This is because they are measuring the same end-point, and should theoretically be related if they are accurately doing so.

Regardless of which of the two routine oxygenators is used during CPB, it has anecdotally been seen that no clinical difference in anaesthetic depth is observed. However, small differences may be detected by measuring the arterial blood concentration of isoflurane. If a difference exists, it suggests that anaesthetists should take the oxygenator transfer characteristics into account when deciding on which isoflurane concentration is to be used. If no difference is established, it will reassure anaesthetists that their interpretation of depth of anaesthesia in the clinical environment is correct.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* who have given their consent to participate
* scheduled for elective cardiac surgery requiring CPB

Exclusion Criteria:• younger than 18 years' old

* unwilling or unable to provide informed consent
* presenting for emergency surgery
* undergoing cardiac surgery without CPB
* in whom total intravenous anaesthesia (TIVA) is being used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2017-04-26 (Actual); Study Completion 2017-04-26 (Actual)

PRIMARY OUTCOMES:
Arterial blood concentration of isoflurane | Application of aortic cross clamp, 20 minutes after application, removal of aortic cross clamp.
  6ml sample of blood will be taken at three time points during an operation requiring cardiopulmonary bypass. This blood will be analysed using gas chromatography and mass spectrometry in order to quantify isoflurane concentrations.
  Mean values will be calculated for each participant, and then an overall mean will be produced for each oxygenator. This will then be compared using independent-samples t-test.

SECONDARY OUTCOMES:
Change in Bispectral Index Score (BIS) | Application of aortic cross clamp, 20 minutes after application, removal of aortic cross clamp.
  A five-electrode BIS monitor will be placed on the forehead at the beginning of surgery. This will display a BIS Score on the Mindray monitor.
Change in arterial temperature | Application of aortic cross clamp, 20 minutes after application, removal of aortic cross clamp.
  Arterial temperature is measured by the cardiopulmonary bypass machine and displayed continuously on the perfusionist's monitors. It will be read directly from these monitors.
Change in exhaust isoflurane concentration | Application of aortic cross clamp, 20 minutes after application, removal of aortic cross clamp.
  The cardiopulmonary bypass exhaust output will be analysed by infrared gas analysis, which will be displayed as a reading on the Mindray monitor throughout the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Alston, Principal Investigator — Honorary Clinical Senior Lecturer and Consultant Anaesthetist
Locations (1):
- Royal Infirmary Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No